CLINICAL TRIAL: NCT04664088
Title: The Efficacy and Safety of Acupuncture for Prophylaxis of Vestibular Migraine
Brief Title: Acupuncture for Prophylaxis of Vestibular Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Principal Investigator, Tianye Hu, doctor, Affiliated Hospital of Jiaxing University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021ZQ084
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Vestibular Migraine
Keywords: vestibular migraine; randomized controlled trial; acupuncture
MeSH Terms: interventions — Acupuncture Therapy; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): Patients in this group will receive acupuncture once every other day (3 days per week) over an 8-week period (a total of 24 sessions).
  Interventions: Procedure: Acupuncture
- Medication group (Active Comparator): Participants in this group will receive oral administration of venlafaxine 50 mg once a day for 8 weeks.
  Interventions: Drug: Venlafaxine

INTERVENTIONS:
Procedure: Acupuncture — Patients in this group will receive acupuncture once every other day (3 days per week) over an 8-week period (a total of 24 sessions). In each session, needles will be retained for 30 minutes. The acupoints will include Baihui (DU20), Qianding (DU21), Houding (DU19), Yintang (DU29), Fengchi (GB20), Shuaigu (GB8), Tongli (HT5), Hegu (LI4), Taichong (LR3), Fenglong (ST40), Xuanzhong (GB39) and Zulinqi (GB41). The selection of acupoints is on the basis of meridian theory and patients' clinical symptoms.
  Patients are not allowed to take prophylactic medications. But in case of intolerable acute VM attacks, the patients will be instructed to take triptans as rescue medication, and the dosage of medication will be documented in the patient diary.
  Arms: Acupuncture group
Drug: Venlafaxine — Participants in this group will receive oral administration of venlafaxine 50 mg once a day for 8 weeks. In case of intolerable acute VM attacks, the patients will be instructed to take triptans as rescue medication, and the dosage of medication will be documented.
  Arms: Medication group

SUMMARY:
With its high incidence rate and low diagnosis rate, vestibular migraine (VM) can seriously affect patients' quality of life. Current treatment of VM mainly contain rescue treatment and prophylaxis, both of which are often pharmacological-based therapies and bring a series of unavoidable side effects, which leads to poor compliance of patients. Moreover, frequent VM attacks can seriously affect patients' daily life and work. Therefore, prophylaxis treatment is of great significance for VM patients. As a non-pharmarceutical therapy, acupuncture is widely used for a wide range of migrainous and emotional disorders. Thus, it might be an alternative treatment for VM, but current evidence remains inconclusive. The aim of this randomized controlled trial is to investigate the prophylactic efficacy and safety of acupuncture therapy in patients with VM.

DETAILED DESCRIPTION:
This randomized controlled trial will enroll patients with vestibular migraine from the First Affiliated Hospital of Jiaxing University. All participants will be randomly assigned to two groups. Participants will receive acupuncture in the treatment group, while participants in the control group will be treated by venlafaxine. All treatments will be given for 8 weeks. The primary outcome measures are change in vertigo/migraine days and vertigo/migraine attacks, vertigo severity, and migraine intensity per 4 weeks from baseline. The secondary outcome measures are change in dosage of rescue medication, anxiety level，depression level，and quality of life per 4 weeks from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age 18 to 80 , male or female;
2. Patients meet the criteria proposed by the collaboration of Barany Society and the International Headache Society in 2012;
3. Vertigo/migraine attacks at least 3 times per month in the last 3 months; or vertigo/migraine days are at least 4 days per month;
4. Patients have unsatisfactory response to rescue treatments and seek for preventive treatments;
5. Patients can fully understand the study protocol and agree to sign written informed consent forms.

Exclusion Criteria:

1. Patients'vertigo and headache are caused by other diseases, such as vestibular neuritis, Meniere disease, tension headache, and other cerebrovascular diseases.
2. Patients have prophylactic headache treatment with drugs in the past 3 months.
3. Patients are receiving adjunctive therapy that is not widely accepted for treating VM, such as Chinese herbs.
4. Patients have severe complications in cardiovascular, cerebrovascular, liver, kidney, hematopoietic and other systems that are not controlled significantly;
5. Pregnant and lactating female patients;
6. Patients have mental illness that affects cognitive function.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of vertigo/migraine days and vertigo/migraine attacks | 4 weeks before intervention, at 4, 8 weeks after intervention and at 4, 8, 16 weeks of follow-up
  The number of vertigo/migraine days and vertigo/migraine attacks will be assessed by a patient diary.
Change in vertigo severity | 4 weeks before intervention, at 4, 8 weeks after intervention and at 4, 8, 16 weeks of follow-up
  Vertigo severity will be measured by dizziness handicap inventory (DHI)
Change in migraine intensity | 4 weeks before intervention, at 4, 8 weeks after intervention and at 4, 8, 16 weeks of follow-up
  Migraine intensity will be measured by visual analogue scale (VAS)

SECONDARY OUTCOMES:
Change in doses of rescue medication | 4 weeks before intervention, at 4, 8 weeks after intervention and at 4, 8, 16 weeks of follow-up
  Doses of rescue medication (triptans) will be documented by patients in the patient diary.
Change in anxiety level | 4 weeks before intervention, at 4, 8 weeks after intervention and at 4, 8, 16 weeks of follow-up
  Anxiety level will be measured by Generalized Anxiety Disorder-7 (GAD-7) scale.
Change in depression level | 4 weeks before intervention, at 4, 8 weeks after intervention and at 4, 8, 16 weeks of follow-up
  Depression level will be measured by Patient Health Questionnaire (PHQ-9) scale
Change in quality of life | 4 weeks before intervention, at 4, 8 weeks after intervention and at 4, 8, 16 weeks of follow-up
  Quality of life will be measure by 36-item short form health survey (SF-36).

CONTACTS AND LOCATIONS:
Overall Officials: Tianye Hu, MM, Principal Investigator — Affiliated Hospital of Jiaxing University
Locations (1):
- The First Affiliated Hospital of Jiaxing University, Jiaxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beh SC. Vestibular Migraine: How to Sort it Out and What to Do About it. J Neuroophthalmol. 2019 Jun;39(2):208-219. doi: 10.1097/WNO.0000000000000791. PMID 31094996
- [Background] Bednarczuk NF, Bonsu A, Ortega MC, Fluri AS, Chan J, Rust H, de Melo F, Sharif M, Seemungal BM, Golding JF, Kaski D, Bronstein AM, Arshad Q. Abnormal visuo-vestibular interactions in vestibular migraine: a cross sectional study. Brain. 2019 Mar 1;142(3):606-616. doi: 10.1093/brain/awy355. PMID 30759189
- [Background] Tedeschi G, Russo A, Conte F, Laura M, Tessitore A. Vestibular migraine pathophysiology: insights from structural and functional neuroimaging. Neurol Sci. 2015 May;36 Suppl 1:37-40. doi: 10.1007/s10072-015-2161-x. PMID 26017509
- [Background] Morganti LO, Salmito MC, Duarte JA, Bezerra KC, Simoes JC, Gananca FF. Vestibular migraine: clinical and epidemiological aspects. Braz J Otorhinolaryngol. 2016 Jul-Aug;82(4):397-402. doi: 10.1016/j.bjorl.2015.06.003. Epub 2015 Oct 29. PMID 26614042
- [Background] Nowaczewska M. Vestibular migraine - an underdiagnosed cause of vertigo. Diagnosis and treatment. Neurol Neurochir Pol. 2020;54(2):106-115. doi: 10.5603/PJNNS.a2020.0031. Epub 2020 Apr 14. PMID 32285435